CLINICAL TRIAL: NCT06446882
Title: Diagnostic HER2DX-guided Treatment for patIents wIth Early-stage HER2-positive Breast Cancer
Acronym: DEFINITIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Clinic Barcelona (Other)
Collaborators: SOLTI Breast Cancer Research Group (Other); Austrian Breast & Colorectal Cancer Study Group (Network); UNICANCER (Other); Westdeutsche Studiengruppe GmbH (WSG) (Unknown); Istituto Oncologico Veneto IRCCS (Other); University College Cork (Other); University of Padova (Other); Istituto Europeo di Oncologia (Other); National University of Ireland, Galway, Ireland (Other); The Sheba Fund for Health Services and Research (Unknown); Erasmus University Rotterdam (Other); Medical University of Vienna (Other); Institut Català d'Oncologia (Other); Europa Donna (Unknown); Reveal Genomics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HCB-ONC002
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: HER2-positive Breast Cancer; Early-stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Treatment by physician´s choice without the diagnostic test results (Other): Treatment by physician´s choice, blinded to the diagnostic HER2DX test results
  Interventions: Other: Treatment by physician´s choice, blinded to the diagnostic HER2DX test results
- Arm B: Personalized treatment according to molecular diagnosis with HER2DX (Experimental): Personalized treatment according to molecular diagnosis with non-blinded HER2DX results
  Interventions: Device: Personalized treatment according to molecular diagnosis with HER2DX

INTERVENTIONS:
Device: Personalized treatment according to molecular diagnosis with HER2DX — Patients with HER2DX high-risk disease:
  * Neoadjuvant treatment:
    * High HER2DX pCR score: paclitaxel per 12 weeks + trastuzumab +/- pertuzumab per 4-5 cycles.
    * Medium HER2DX pCR score: carboplatin + paclitaxel per 12-18 (or docetaxel per 4-6 cycles) + trastuzumab +/- pertuzumab per 4-7 cycles.
    * Low HER2DX pCR score: standard of care neoadjuvant CT regimens and HER2 blockade at the investigator's choice.
  * Adjuvant treatment:
    * pCR at surgery; Trastuzumab +/- pertuzumab up to a total of 18 cycles (including neoadjuvant and adjuvant therapy).
    * No pCR at surgery: T-DM1 per 14 cycles.
  Patients with HER2DX low-risk disease:
  * Neoadjuvant treatment: paclitaxel per 12 weeks + trastuzumab +/- pertuzumab per 4-5 cycles.
  * Adjuvant treatment will be according to the pCR status at surgery:
    * pCR at surgery: trastuzumab or no adjuvant treatment.
    * No pCR at surgery: trastuzumab or T-DM1.
  Arms: Arm B: Personalized treatment according to molecular diagnosis with HER2DX
Other: Treatment by physician´s choice, blinded to the diagnostic HER2DX test results — Patients randomized in ARM A will be treated with standard of care neoadjuvant CT regimens and HER2 blockade at the investigator's choice validated by national and/or international guidelines.
  Arms: Arm A: Treatment by physician´s choice without the diagnostic test results

SUMMARY:
The primary goal of the DEFINITIVE trial is to demonstrate the effectiveness of the HER2DX diagnostic assay in enhancing the management of patients with early-stage HER2- positive breast cancer.

Patients randomized to arm A will receive adjuvant treatment by physician´s choice, blinded to the diagnostic HER2DX test results. Patients randomized to Arm B will receive personalized treatment according to HER2DX results.

DETAILED DESCRIPTION:
This is an international, multicenter, prospective, randomized, two-arm, open-label, phase III study to evaluate the HRQoL, safety, efficacy, and economical costs of using HER2DX in patients with stage II to IIIA HER2-positive breast cancer, suitable for neoadjuvant therapy.

A dual primary endpoint with an according multiple testing procedure is defined in this study. First, the study will evaluate superiority in quality of life using i) the GHS scale from the EORTC QLQ-C30 questionnaire version 3.0 and ii) the score from the FACIT Fatigue Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to any trial-specific procedure. Note: Candidate patients in France must be affiliated to a Social Security System (or equivalent).
2. Male/female patients who are at least 18 years of age on the day of signing informed consent.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Eligible for any of the following drugs: taxane, carboplatin, trastuzumab, pertuzumab and T-DM1 therapy.
5. Histologically confirmed non-metastatic primary invasive adenocarcinoma of the breast untreated and recently diagnosed.
6. Stage at presentation: cT1 cN1-2 or cT2-3 cN0-2 as determined by AJCC staging system, 8th edition (specifically in accordance with Anatomic Stage group rules).

   Note: Axillary lymph node status must be assessed by fine needle biopsy or core biopsy. This procedure at screening will be omitted if there is no suspicion for positive axillary lymph node(s) radiographically or if a pathological report of suspicious lymph nodes of the results of a fine needle biopsy or core biopsy is available prior to the screening period.
7. Absence of distant metastasis (i.e., cM0).
8. Patients with multifocal tumors (more than one mass confined to the same quadrant as primary tumor) are eligible provided at least one focus is sampled and locally confirmed as HER2-positive.
9. Patients with multicentric tumors (multiple tumors involving more than one quadrant) are eligible provided all discrete lesions are sampled and locally confirmed as HER2-positive.

   Note: In patients with multifocal or multicentric breast cancer, the largest lesion should be measured to determine T stage and to performe the HER2DX test.
10. HER2 positivity defined as either of the following: IHC 3+ or HER2 2+/ ISH positive as per most recent ASCO- CAP guideline according to the local laboratory as determined on the most recently analyzed tissue sample.
11. ER/PR status determined local based on pretreatment breast biopsy material according to the most recent ASCO/CAP guidelines.
12. Candidates for neoadjuvant treatment.
13. Patient agreement to undergo appropriate surgical management, including axillary lymph node surgery and partial or total mastectomy, after completion of neoadjuvant treatment
14. Baseline left ventricular ejection fraction (LVEF) ≥ 50% measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scans.
15. Availability of pre-treatment tumor tissue sample of FFPE tumor block from primary tumor in the breast for diagnostic HER2DX test. The tumor tissue should be of good quality based on total and viable tumor content and must be evaluated centrally for quality prior to enrollment. Archival tumor tissue or ex professo biopsy are acceptable.
16. Adequate hematologic and end-organ function.
17. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs, as defined below:

    * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period, 6 months after the final dose of doxorubicin, 12 months after the final dose of cyclophosphamide, 6 months after the final dose of paclitaxel, and 7 months after the final dose of trastuzumab, pertuzumab, or T-DM1, whichever occurs last. Women must refrain from donating eggs during this same period.
    * A woman is of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (> 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
    * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, copper intrauterine devices, hormonal contraceptives that inhibit ovulation, and hormone-releasing intrauterine devices in women with hormone receptor-negative tumors only; the use of hormonal contraceptives and hormone releasing intrauterine devices are prohibited in women with hormone receptor-positive tumors.
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
18. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

    * With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 6 months after the final dose of doxorubicin and/or cyclophosphamide, 6 months after the final dose of paclitaxel, and 7 months after the final dose of trastuzumab, pertuzumab, or T-DM1, whichever occurs last. Men must refrain from donating sperm during this same period. Male patients are encouraged to seek advice regarding cryoconservation of sperm prior to commencing study treatment because of the possibility of infertility with CT.
    * With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of doxorubicin and/or cyclophosphamide, 6 months after the final dose of paclitaxel, and 7 months after the final dose of trastuzumab, pertuzumab, or T-DM1, whichever occurs last to avoid exposing the embryo.
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer.
2. Known hypersensitivity to any of the excipients of trastuzumab, pertuzumab, carboplatin, T-DM1, docetaxel or paclitaxel.
3. Patients with synchronous bilateral invasive breast cancer.
4. Prior systemic therapy for treatment of breast cancer.
5. Ulcerating or inflammatory breast cancer.
6. Undergone incisional and/or excisional biopsy of primary tumor and/or axillary lymph nodes.
7. Sentinel lymph node procedure or axillary lymph node dissection prior to initiation of neoadjuvant therapy.
8. Patients with a history of previous breast cancer are excluded. Patients with a history of any other cancers (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years are excluded. For patients with a history of other non-breast cancerscancerscancers within 3 years and considered of low risk of recurrence per investigator's judgment (for example, papillary thyroid cancer treated with surgery), eligibility is to be discussed with the Sponsor.
9. Cardiopulmonary dysfunction as defined by any of the following prior to randomization:

   * History of congestive heart failure of any classification.
   * Angina pectoris requiring anti-anginal medication, serious cardiac arrhythmia not controlled by adequate medication, severe conduction abnormality, or clinically significant valvular disease.
   * High-risk uncontrolled arrhythmias (i.e., atrial tachycardia with a heart rate > 100/min at rest, significant ventricular arrhythmia [ventricular tachycardia], or higher-grade atrioventricular [AV]-block [second degree AV-block Type 2 [Mobitz 2] or third-degree AV-block]).
   * Significant symptoms (Grade > 1) relating to left ventricular dysfunction, cardiac arrhythmia, or cardiac ischemia.
   * Myocardial infarction within 12 months prior to randomization.
   * Evidence of transmural infarction on ECG.
   * Requirement for oxygen therapy.
   * Dyspnea at rest.
10. Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment or anticipation of need for a major surgical procedure during the Study.
11. Severe infection within 4 weeks prior to initiation of Study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
12. History of significant co-morbidities that, in the judgment of the investigator, may interfere with the conduction of the Study, the evaluation of response, or with consent procedure.
13. Pregnancy or breastfeeding, or intention of becoming pregnant during Study treatment or within 6 months after the final dose of paclitaxel, or 7 months after the final dose of trastuzumab, pertuzumab, or T-DM1, whichever occurs last.

    Note: Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of Study treatment.
14. Persons deprived of their liberty or under protective custody or guardianship.
15. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial, social, or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Global health status (GHS) scale from the EORTC QLQ-C30 questionnaire | Up to 5 years
  The GHS scale is based on two 7-point questions (from very poor to excellent, items 29-30 from EORTC QLQ-C30 questionnaire).
  Following EORTC scoring manuals, a linear transformation will be used to standardize the GHS scale to a 0-100 scale.
Score from the FACIT Fatigue Scale | Up to 5 years
  The FACIT Fatigue Scale, version 4 will be used to evaluate PRO measures of quality-of-life concerns related to fatigue.
  The FACIT Fatigue Scale is a 13-item questionnaire designed to measure fatigue and its impact on daily life in individuals with various health conditions. Respondents rate their fatigue experiences over the past week on a scale from 0 to 4, with higher scores indicating less fatigue. The total score ranges from 0 to 52.

SECONDARY OUTCOMES:
Functional and symptom scales from the EORTC QLQ-C30 questionnaire. | Up to 5 years
  Change from baseline in all other functional and symptom scales (items 1 to 28) from the EORTC QLQ-C30 questionnaire version 3.0 to assesses cancer-related symptoms, impacts, and treatment-related symptoms.
  The items are rated on a 4-point rating scale ranging from 0 ("not at all") to 4 ("very much").
Score of the EuroQol-5D | Up to 5 years
  Change from baseline in the score of the EuroQol-5D.
  The 5-level version EQ-5D-5L is a 6-item generic patient-reported preference-based instrument designed to assess health status of patients. The EQ-5D-5L consists of 2 sections:
  * the EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels of severity: the dimensions of mobility, self-care, and usual activity are rated ranging from 1 (no problem completing task) to 5 (unable to complete task) while the dimensions of pain/discomfort and anxiety/depression are rated ranging 1 (no symptom) to 5 (extreme symptom).
  * the EuroQoL visual analogue scale (EQ-VAS) is for patients to self-rate their (global) health state utilizing a vertically oriented visual analogue scale where 100 represents the "best possible health state" and 0 represents the "worst possible health state".
pCR rates | Up to 5 years
  pCR rates between groups at randomization and according to the predefined HER2DX pCR score as a continuous variable and as group categories.
  pCR will be defined as the complete absence of invasive carcinoma in the breast and axillary lymph nodes on histological examination at the time of definitive surgery, irrespective of in situ carcinoma in the breast.
Residual cancer burden (RCB) | Up to 5 years
  RCB between groups at randomization and according to HER2DX pCR score as a continuous variable and as group categories.
  Residual cancer burden (RCB) is defined as classes 0, 1, 2 and 3, according to the MD Anderson Cancer Center recommendations by local evaluation.
Invasive disease-free survival (iDFS) | Up to 5 years
  Invasive disease-free survival (iDFS) between groups at randomization and according to HER2DX pCR score in continuous variable and risk group.
  iDFS is defined as the time from surgery until the date of the first occurrence of one of the following events: recurrence of ipsilateral invasive breast tumor, recurrence of ipsilateral locoregional invasive disease, a distant disease recurrence, contralateral invasive breast cancer, second primary or death from any cause.
Distant metastasis free survival (DMFS) | Up to 5 years
  Distant metastasis free survival (DMFS) between groups at randomization and according to HER2DX pCR score in continuous variable and risk group.
  DMFS is defined as the time from surgery to date of first event of distant metastatic recurrence or death (any cause). Contralateral breast cancer and secondary cancers will not be considered. Patients who do not have a DMFS event will be censored at the last recurrence assessment. Patients alive with no evidence of metastasis at the time of their last visit are censored at the time of the last examination.
Recurrence-free interval (RFI) | Up to 5 years
  Recurrence-free interval (RFI) between groups at randomization and according to HER2DX pCR score in continuous variable and risk group.
  RFI is defined as from surgery until the date of the first occurrence of one of the following events: recurrence of ipsilateral breast tumor (in situ or invasive), recurrence of ipsilateral locoregional invasive disease, a distant disease recurrence, contralateral invasive breast cancer or death from breast cancer.
Event free survival (EFS) | Up to 5 years
  Event free survival (EFS) between groups at randomization and according to HER2DX pCR score in continuous variable and risk group.
  EFS is defined as the time from randomization to the first documented disease recurrence, unequivocal tumor progression determined by the treating investigator, or death from any cause, whichever occurs first.
Incidence, duration, and severity of adverse events (safety and tolerability) | Up to 5 years
  Incidence, duration, and severity of adverse events (AEs) assessed by the NCI Common Terminology for Classification of AEs (CTCAE) version 5, including dose reductions, delays, and treatment discontinuations.
CAHPS cancer care survey (AHQR) | Up to 5 years
  Patient-reported Experience Measurement (PREM) data will be elicited from the patients in this study to fully understand the experience of patient.
  Team accessibility, Communication, Information from care providers, Care continuum coordination, respect and courtesy, secondary effects management, shared-decision making, language barriers and overall care perception, will be evaluated using the Drug Therapy Team survey and the Supplementary Items survey from the CAHPS cancer care survey (AHQR).
  The Drug Therapy Team Survey is a 56 items questionnaire designed to measure accessibility to the care team, quality of information provided, quality of the visit, management of the impact of the disease on daily life, quality of the administration staff support, and a global scale from 0 to 10 to rate the quality of the team.
  The supplementary items survey is a 16 items questionnaire and measure three dimensions of experience: access, information and shared-decision making.
Economic impact of the HER2DX test | Up to 5 years
  Health economic evaluation to analyse the cost-effectiveness in patients with and without HER2DX test information, not only direct cost for hospitals/public health system, but also indirect cost from a societal perspective.
  The EuroQol-5D-5L questionnaire will be used to calculate a health status utility score for use in health economic analyses.
Work productivity | Up to 5 years
  To evaluate whether the potential treatment de-escalation following tailored treatment by HER2DX could have impact in the work productivity using the Work Productivity and Activity Impairment Questionnaire (WPAI- GH).The WPAI-GH is a 6-item instrument that gauges absenteeism (missed work time due to the health issue), presenteeism (decreased productivity while working due to the health problem), overall work hindrance, and limitations in daily activities.

CONTACTS AND LOCATIONS:
Locations (15):
- Austria (4):
  - Lkh Hochsteiermark-Leoben, Leoben
  - Ordensklinikum Linz, Barmherzige Schwestern, Bhs, Linz
  - Uniklinikum Salzburg, Salzburg
  - Klinikum Wels-Grieskirchner, Wels
- Sheba Medical Center, Ramat Gan, Israel
- Spain (10):
  - Instituto Catalán de Oncología (ICO) - Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Clínico San Cecilio, Granada, Granada
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, La Coruña
  - Complejo Asistencial Universitario de León, León, León
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de Arrixaca, Murcia, Murcia
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Instituto Catalán de Oncología (ICO) - Badalona, Badalona
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No